CLINICAL TRIAL: NCT04906525
Title: Effects of 6-week Resistance Training Intervention on Gut Microbiome and Cardiometabolic Outcomes in Adults With Overweight and Obesity
Brief Title: Resistance Training Effects on Gut Microbiome and Cardiometabolic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jaapna Dhillon, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2054484
Record Dates: First submitted 2021-05-05; First posted 2021-05-28 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Exercise Intervention
Keywords: Gut Microbiome; Resistance Training; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical activity guidelines (Other): Participants are given recommendations on physical activity guidelines
  Interventions: Other: Conventional physical activity guidelines
- Resistance training (Experimental): Participants will undergo 6 weeks of supervised resistance training
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — Participants will undergo 6 weeks of supervised resistance training
  Arms: Resistance training
Other: Conventional physical activity guidelines — Participants are given recommendations on physical activity guidelines
  Arms: Conventional physical activity guidelines

SUMMARY:
The overall objective of this study is to investigate the effects of resistance training on the gut microbiome and cardiometabolic outcomes in adults with overweight and obesity.

DETAILED DESCRIPTION:
The overall objective of this study is to investigate the effects of resistance training on the gut microbiome and cardiometabolic outcomes in adults with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* BMI: 25-45 kg/m2
* Sedentary lifestyle
* Consistent diet patterns
* Weight-stable (<4 kg change over the last 3 mo)
* Willingness to adhere to resistance training protocol and not change diet
* Non-smoker >1 year or more

Exclusion Criteria:

* Disabilities preventing adherence to resistance training protocol
* Recent start of medications that affect metabolism or appetite
* Antibiotics
* Diabetes
* Drug therapy for coronary artery disease, peripheral artery disease, congestive heart failure, or dyslipidemia
* Uncontrolled hypertension and blood pressure ≥ 180/110
* Gastrointestinal disease and/or bariatric surgery
* Smoking
* Illicit drug use
* Pregnant or lactating individuals

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in stool microbiome diversity | Change over 6 weeks
  16s rRNA sequencing
Change in stool microbiome composition | Change over 6 weeks
  16s rRNA sequencing

SECONDARY OUTCOMES:
Change in blood pressure | change over 6 weeks
  diastolic and systolic blood pressure
Fat mass | Change over 6 weeks
  body composition
Fat free mass | Change over 6 weeks
  body composition
Change in fasting glucose | change over 6 weeks
  Fasting Glucose
Change in glucose regulation | change over 6 weeks
  2 hour glucose clearance
Hip circumference | change over 6 weeks
  anthropometrics
Waist circumference | change over 6 weeks
  anthropometrics
Physical activity | change over 6 weeks
  kcalories burned during free living activity measured by accelerometer
Sleep Quality | change over 6 weeks
  Measured using actigraphs
Sleep Duration | change over 6 weeks
  Measured using actigraphs
24hr appetite ratings | Once at baseline and at the end of 6 week intervention
  Subjective rating using visual analog scales
Change in Body mass | change over 6 weeks
  Measured in kg
Short chain fatty acids | Change over 6 weeks
  Acetate, propionate, and butyrate

OTHER OUTCOMES:
Food environment perceptions | baseline and at the end of 6 week intervention
  subjective and objective questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jaapna Dhillon, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported here after deidentification (text, tables, figures, etc.)
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be deposited in online data repositories.